CLINICAL TRIAL: NCT05827133
Title: A Non-Interventional Study to Evaluate the Effect of Intraocular Lens (IOL) Centration and Tilt on Visual Performance in Patients Who Have Undergone Clareon® Vivity® IOL Implantation
Brief Title: Effect of Intraocular Lens (IOL) Centration and Tilt on Visual Performance With Clareon® Vivity® IOL Implantation
Status: Completed | Type: Observational
Sponsor: East Coast Institute for Research (Network)
Collaborators: Alcon Research (Industry); Florida Eye Specialists (Unknown)
Responsible Party: Sponsor
Other Study IDs: ECIR-Alcon-01
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cataract; Lenses, Intraocular
Keywords: Extended Depth of Focus Lens; Toric Lens; Decentration; Tilt; Clareon Vivity; Clareon Vivity Toric
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Individuals implanted with Clareon® Vivity® or Vivity® Toric Intraocular Lenses (IOLs)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to assess the effect of intraocular lens (IOL) movement in patients who have undergone Clareon® Vivity® IOL implantation.

The main question it aims to answer is: Does an association exist between IOL movement and patient quality of vision?

Participants implanted with Clareon® Vivity® and Vivity® Toric IOLs will be asked to do the following:

* consent to participate in the study
* allow researchers to access their personal medical records
* undergo a series of tests to assess the position of their IOLs and quality of vision

Researchers will assess participant examination results to determine whether an association exists between IOL movement and patient quality of vision.

DETAILED DESCRIPTION:
This is a non-interventional, single-center, multi-surgeon, observational study to evaluate the effect of intraocular lens (IOL) centration and tilt on visual performance in patients who have undergone Clareon® Vivity® IOL implantation. The study population will include individuals implanted with Clareon® Vivity® and Vivity® Toric IOLs. IOL implantations reviewed will range from the earliest performed (May 2022) onward, until 100 implanted patients (200 eyes) are enrolled. Potential subjects will be consented, then retrospective chart review of pre-operative and operative implantation data will occur and postoperative data will be collected (1 or more months post-operation) via examination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* History of adult cataract and uneventful, refractive cataract surgery with Clareon® Vivity® or Vivity® Toric intraocular lens (IOL) implantation with manifest refraction spherical equivalent (MRSE) within ±1.00 D
* Willing to undergo an eye exam with pupil dilation

Exclusion Criteria:

* Moderate to severe posterior capsule opacification (2+ or more)
* Yttrium aluminum garnet (YAG) laser capsulotomy within 1 month prior to enrollment
* Laser-assisted in situ keratomileusis (LASIK) or photorefractive keratectomy (PRK) within the one year prior to IOL implantation or any time after IOL implantation
* Any previous ocular surgery (excluding YAG, LASIK, PRK)
* Clinically significant ocular pathology; severe diabetic retinopathy, age-related macular degeneration (AMD), glaucoma, severe dry eye, irregular astigmatism, zonular weakness, pseudoexfoliation, ocular trauma
* Any additional procedure(s) at the same time as the Vivity implantation including but not limited to microinvasive glaucoma surgery (MIGS)
* Women who are pregnant at the time of screening (based on self-reported history)
* Medical or other problems which in the opinion of the investigator will render study participation unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include approximately 100 adult participants (200 eyes) who have previously been implanted with Clareon® Vivity® and Vivity® Toric intraocular lenses (IOLs).
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Monocular best-corrected distance visual acuity (BCDVA) (4 m) (logMAR) | Visit 1

SECONDARY OUTCOMES:
Decentration of intraocular lens (IOL) (mm) | Visit 1
Tilt of intraocular lens (IOL) (°) | Visit 1
Monocular uncorrected distance visual acuity (UCDVA) (4 m) (logMAR) | Visit 1
Monocular distance-corrected intermediate visual acuity (DCIVA) (66 cm) (logMAR) | Visit 1
Monocular uncorrected intermediate visual acuity (UCIVA) (66 cm) (logMAR) | Visit 1
Manifest refraction/Manifest refraction spherical equivalent (MRSE) (D) | Visit 1

OTHER OUTCOMES:
Mean photopic low contrast (25%) monocular best-corrected distance visual acuity (BDCVA) (4 m) (logMAR) | Visit 1
Mesopic pupil size (mm) | Visit 1
Coma higher-order aberration (HOA) (µm) | Visit 1
Spherical higher-order aberration (HOA) (µm) | Visit 1

CONTACTS AND LOCATIONS:
Locations (1):
- East Coast Institute for Research, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No